CLINICAL TRIAL: NCT05778175
Title: Common Cases in Pediatric Intensive Care in Assuit University Cardiology Institute, a Clinical Audit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Tharwat Attia salama, Resident Doctor, Assiut University
Other Study IDs: Clinical audit on Cardiac ICU
Record Dates: First submitted 2023-03-05; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Congenital Heart Disease in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1Evaluation of the management methods according to guidelines for cardiac patients admitted to Intensive care in pediatric Assuit university cardiology institute and the effectiveness and outcome of following of these medications comparing them with international advanced centers.

Types of shocks in cardiac patients and management of cardiogenic shock needs especial concern.

DETAILED DESCRIPTION:
Critically ill pediatric patients with cardiac disease such as (cardiogenic Shock, life- threatening arrhythmias, congenital heart diseases with unstable cardiorespiratory status, uncompensated heart failure, after cardiac catheterization and after high risk cardiovascular and intrathoracic procedures) must be admitted to a designated intensive care unit and not discharged untill reversal of the disease process or restoration of the unstable physiologic condition and become hemodynamically stable, cardiac dysrhythmias controlled and there's no need for intravenous inotropic support, vasodilators, and antiarrhythmic drugs or when required, low doses of these medications can be administered safely .

Physicians, nurses and other health care providers should perform a regular review of their clinical practice and the activities which carried out relying on established standards and the main purpose of this revision process is to evaluate the efficacy, effectiveness and safety of the provided medical care .

Because the number of patients with critical heart diseases is relatively small, there are big knowledge gaps and variation in the methods of management. Presence of a specific Pediatric Cardiac Intensive Care led to correction of this knowledge gap and providing clinicians with Scientific statements and white papers used as a guidance in diagnostic and therapeutic strategies aiming to changing the individual institution-based practices efforts to national standardized protocols which results in a better outcome .

Presence of a specific cardiac intensive care unit (CICU) with highly specialized teams with specific knowledge and skills leads to direction of many investigations to provide the highest value care. This has many advantages on the outcome of the admitted patients such as: lower hospital costs, shorter duration of hospital stay and decrease mortality rate .

A case of special concern is cardiogenic shock which is an acute state of circulatory failure due to impairment of myocardial contractility and it's the most serious stage of heart failure and a major cause of morbidity and mortality in pediatric cardiac patients, it must be recognized and managed early and any delay in the recognition and management of potential clinical symptoms and signs of compensated shock could lead to a high mortality rate .

Recognition of early signs of cardiogenic shock by clinical examination (tachycardia, hypotension, impaired conscious level, fall in oxygen saturation, decreased urine output and respiratory distress) or investigations like as: chest x-ray (cardiomegaly, pulmonary edema), ECG (arrhythmias, conduction disorders, myocardial ischemia),and transthoracic echocardiograms are useful for diagnostic, etiological, therapeutic, and prognostic purposes .

Initial management of the cardiogenic shock aiming to restore adequate oxygen delivery to peripheral tissues by oxygen therapy (noninvasive or invasive ventilation) with a saturation objective of >95 % except in cyanotic heart, decrease the circulatory preload by fluid restriction and diuretics, decrease the circulatory afterload by arterial vasodilators, increase the cardiac contractility by inotropes (dopamine, dobutamine and digoxin) and treating curable causes (fluid and electrolyte balance, rhythm, or thromboembolic disorders; pneumothorax, tamponade, infection) .

ELIGIBILITY:
Inclusion Criteria:

* All cardiac patients aged from 30 days to 18 years old admitted in the pediatric intensive care Assuit University cardiology Institute within one year

Exclusion Criteria:

* Other pediatric cardiac patient admitted in the cardiology unit outside the Intensive care.

Ages: 30 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Observational study on the methods of management of the common cases in pediatric cardiac intensive care
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Common cases in Pediatric Intensive care in Assuit University Cardiology Institute, a clinical audit | Baseline
  Evaluation of different methods of management and comparing them with the guidelines of diagnosis and treatment aiming to changing the individual institution-based practices efforts to national standardized protocols which results in a better outcome by a questionnaire.

REFERENCES:
- [Background] Guidelines for the transfer of critically ill patients. Guidelines Committee of the American College of Critical Care Medicine; Society of Critical Care Medicine and American Association of Critical-Care Nurses Transfer Guidelines Task Force. Crit Care Med. 1993 Jun;21(6):931-7. PMID 8080468
- [Background] Reddy S, Polito A, Staveski S, Dalton H. A process for academic societies to develop scientific statements and white papers: experience of the Pediatric Cardiac Intensive Care Society. Cardiol Young. 2019 Feb;29(2):174-177. doi: 10.1017/S1047951118002019. Epub 2018 Dec 4. PMID 30511598